CLINICAL TRIAL: NCT02422498
Title: A Phase II Trial of Homologous Recombination Repair Status as a Biomarker of Response in Locally Recurrent/Metastatic Triple Negative Breast Cancer Patients Treated With Concurrent Cisplatin and Radiation Therapy
Brief Title: Homologous Recombination Repair Status as a Biomarker of Response in Locally Recurrent/Metastatic Triple Negative Breast Cancer Patients Treated With Concurrent Cisplatin and Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Cedars-Sinai Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-032
Record Dates: First submitted 2015-04-14; First posted 2015-04-21 (Estimated); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2022-12

CONDITIONS: Locally Recurrent/Metastatic Triple Negative Breast Cancer
Keywords: Treated with Concurrent Cisplatin; Treated with Radiation Therapy; Homologous Recombination Repair Status; Biomarker of Response; 15-032; Patients
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Cisplatin

ARMS (1):
- Concurrent Cisplatin & Radiation Therapy (Experimental)
  Interventions: Radiation: external beam radiation therapy; Drug: cisplatin; Procedure: Biopsy of Target Tumor

INTERVENTIONS:
Radiation: external beam radiation therapy — Radiation therapy to the target tumor will be delivered with external beam radiation therapy. In metastatic cases where the intent is palliative, the dose of radiation will be 3750 cGy delivered in 15 daily fractions, 4-5 days a week. In locoregionally recurrent cases where the intent is to enhance locoregional control, the dose of radiation will be 5000 cGy delivered in 25 fractions, 4-5 days a week plus an optional 10-14 Gy boost to areas of gross tumor.
Drug: cisplatin — Cisplatin treatment should be initiated following study registration. The dose of cisplatin is established as 25 mg/m^2 ivpb once a week (+ 3 days) for 1-2 weeks prior to radiation. The length of one cycle of Cisplatin is 21 days.
Procedure: Biopsy of Target Tumor — Biopsy of the tumor to be irradiated will be performed. Fresh tissue specimens will be sent to the laboratory for performance of the MSK-HRR Assay.

SUMMARY:
The study is being done to find out if the results of a pre-treatment biopsy can predict response to cisplatin and radiation treatment for patients with metastatic or recurrent triple negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed invasive triple negative breast cancer (ER <1%, PR <1%, her-2-neu 0-1+ by IHC or FISH-negative) or as determined by MD discretion
* Radiation to the recurrent or metastatic site is clinically indicated and would be considered standard care for palliation or for locoregional control
* Age ≥18 years
* Tumor to be irradiated is measurable by RECIST 1.1 or PRC
* Willingness to undergo tumor biopsy prior to initiation of treatment
* Life expectancy greater than 6 months
* ECOG performance status 0-2
* Any prior chemotherapy is allowed including prior treatment with platinum-containing chemotherapy
* Prior treatment with FDA-approved or investigational biologics or novel molecularly target therapies, including oral or IV formulations, are permitted.
* Patients must be off prior targeted therapy for at least 14 days prior to study biopsy.
* Use of an effective means of contraception in women of child-bearing potential
* Ability to comprehend and sign informed consent
* Adequate organ and marrow function within 14 days prior to study entry, defined as:

  * Absolute neutrophil count (ANC)>1000/mm3
  * Hemoglobin >9 gm/dl
  * Platelets >100,000/mm3
  * Serum creatinine <1.5 mg/dl OR creatinine clearance of ≥ 50 cc/min
  * SGOT/SGPT<2.5X institutional ULN (<5X ULN if known liver metastases)

Exclusion Criteria:

* Unmeasurable target tumor site by RECIST 1.1 or PRC (ex: lesions <2 cm on CT or MR scan, leptomeningeal disease, ascites, pleural/pericardial effusion, lymphangitis, non-FDG-avid skin lesions)
* Brain metastases requiring focal or whole brain radiation will be excluded, as these lesions cannot be biopsied and can have life expectancies <6 months.
* Inability to obtain a biopsy of the tumor as deemed by the study Interventional Radiologist
* Prior chemotherapy completed <7 days prior to planned study entry
* Prior RT is allowed and must have been completed more than 7 days before planned study entry.

  * Note: For re-irradiation cases, standard departmental guidelines should be followed so as to not exceed normal tissue
* Life expectancy less than 6 months
* Intercurrent illness or other major medical condition or comorbid condition that might affect study participation (uncontrolled renal, pulmonary or hepatic dysfunction or infection)
* Renal dysfunction for which cisplatin dose would be considered unsafe.
* Women on study must be neither pregnant nor nursing nor expected to become pregnant during therapy. For premenopausal women, negative pregnancy test within 14 days of RT is required.
* Concurrent active malignancy other than non-melanomatous skin cancer or carcinoma in-situ of the cervix, unless treatment for the previous cancer was completed >2 years prior to study entry and patient has remained disease-free.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Powell, MD,PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Concurrent Cisplatin & Radiation Therapy
Started | 49
Completed | 45
Not Completed | 4
Not completed — Inevaluable | 4

BASELINE CHARACTERISTICS:
Arm/Group | Concurrent Cisplatin & Radiation Therapy
Number analyzed (Participants) | 49
Age, Continuous [Median (Full Range); unit: years] | 54 [30 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 27
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Response (RECIST 1.1 vs. PET Response Criteria (PRC) as Measurement Tools for Treatment Response)
Description: RECIST 1.1 as measurement tools for treatment response.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent Cisplatin & Radiation Therapy
Number analyzed (Participants) | 49
Participants
  Partial Response | 2
  Progression of Disease | 25
  Not Entered | 22

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Concurrent Cisplatin & Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 40/49
Serious Adverse Events (participants affected / at risk) | 12/49
Other Adverse Events (participants affected / at risk) | 45/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Concurrent Cisplatin & Radiation Therapy (N=49)
Acute kidney injury (Renal and urinary disorders) | 2
Anemia (Blood and lymphatic system disorders) | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Breast infection (Infections and infestations) | 1
Confusion (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Musculoskeletal & conn tissue disorder Other (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 1
Paresthesia (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Skin infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
White blood cell decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Concurrent Cisplatin & Radiation Therapy (N=49)
Fatigue (General disorders) | 25
Anemia (Blood and lymphatic system disorders) | 18
Dermatitis radiation (Injury, poisoning and procedural complications) | 18
Nausea (Gastrointestinal disorders) | 18
White blood cell decreased (Investigations) | 18
Neutrophil count decreased (Investigations) | 16
Lymphocyte count decreased (Investigations) | 13
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Peripheral sensory neuropathy (Nervous system disorders) | 7
Platelet count decreased (Investigations) | 7
Constipation (Gastrointestinal disorders) | 6
Dysgeusia (Nervous system disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 6
Pain (General disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 6
Alanine aminotransferase increased (Investigations) | 5
Dry mouth (Gastrointestinal disorders) | 5
Localized edema (General disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Weight Loss (Investigations) | 5
Dizziness (Nervous system disorders) | 4
Tinnitus (Ear and labyrinth disorders) | 4
Blood and lymphatic system disorders - other (Blood and lymphatic system disorders) | 3
Breast pain (Reproductive system and breast disorders) | 3
Creatinine increased (Investigations) | 3
Edema limbs (General disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT02422498/Prot_SAP_000.pdf